CLINICAL TRIAL: NCT06446934
Title: Continual Optical Cuffless Monitoring to Assess the CPAP Therapeutic Effect on Blood Pressure in Obstructive Sleep Apnea Patients
Brief Title: AKTIIA OBPM to Assess CPAP Effect on Blood Pressure in Obstructive Sleep Apnea
Acronym: AVLA1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Araba (Other)
Collaborators: Bioaraba Health Research Institute (Network)
Responsible Party: Principal Investigator, Mikel Azpiazu, Medical Doctor, Hospital Universitario Araba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS2023034
Record Dates: First submitted 2024-05-27; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Hypertension; Cardiac Function and Hemodynamics; Usability; Patient Experience
Keywords: Hypertension; Obstructive Sleep Apnea; Blood Pressure Monitors; Continuous Positive Airway Pressure; Echocardiography; Pulse Wave Analysis; Photoplethysmography; Telemedicine
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Single-center, single-arm, interventional pre-post design study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPAP (Other): Interventional pre-post CPAP therapy
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — Initial CPAP titration and subsequent CPAP therapy for 12 weeks

SUMMARY:
The goal of this clinical trial is to learn if positive airway pressure (CPAP) therapy works for blood pressure (BP) control in obstructive sleep apnea (OSA) adult patients plus undiagnosed hypertension (HBP), using a cuffless bracelet for continual optical BP monitoring (AKTIIA OBPM).

It will also learn if CPAP improves cardiac function in these patients using speckle tracking echocardiography (STE) and to learn about ease of use and patient experience with AKTIIA device and AKTIIA OBPM.

The main questions it aims to answer are:

* Does CPAP reduce systolic BP (and other BP metrics) in this population?
* Does CPAP improve cardiac function in the same population? Researchers will compare BP metrics derived from AKTIIA OBPM and STE metrics in a before and after CPAP therapy to evaluate its therapeutic effect.

Participants will:

* Take a CPAP titration and telemonitoring program for 12 weeks (from the titration date)
* Take an AKTIIA OBPM one week before CPAP and 12 weeks since CPAP titration date
* Take a STE test twice, before starting CPAP and 12 weeks after CPAP titration date
* Take an online survey about easy of use and patient experience with AKTIIA OBPM device

DETAILED DESCRIPTION:
Patients with moderate-severe OSA, indication for CPAP therapy and undiagnosed hypertension will be included. If the patient meets all the inclusion criteria and none of the exclusion criteria, he/she will be considered a candidate for the study. Once the informed consent has been signed, a visit will be made to initiate continuous blood pressure monitoring with the AKTIIA system (AKTIIA OBPM). The first week (week 0, preCPAP) serves to confirm the presence of HBP (average BP 130/80+ mmHg and/or average nocturnal BP 120/70+ mmHg).

If the participant has HBP criteria, an speckle tracking echocardiography (STE) will be performed (preCPAP) and then CPAP treatment will be initiated following the sleep unit´s telemonitoring care program with initial ambulatory pressure titration. If the participant do not have HBP criteria, only CPAP treatment will be started.

The CPAP titration date will be day 1 for AKTIIA OBPM and CPAP monitoring. At 12 weeks of monitoring, a second STE will be scheduled (post-CPAP) and the end-of-study on-site visit is performed to assess: efficacy and adherence to CPAP, clinical and BP control in the AKTIIA OBPM (week 12, post-CPAP).

Finally, an anonymous electronic survey on AKTIIA device usability and patient experience with AKTIIA OBPM and CPAP therapy will be conducted.

Withdrawal criteria are: ineffective CPAP titration, CPAP dropout, invalid AKTIIA OBPM or dropout, prescription of antihypertensive drug, patient decision or PI decision and loss of contact.

Researchers will compare pre-post CPAP blood pressure metrics (systolic BP as the main parameter), circadian profile, dynamic metrics, STE metrics, efficacy and CPAP adherence, symptoms (ESS, QOL own scales) and subgroup analysis by gender, age, OSA severity or CPAP adherence.

ELIGIBILITY:
Inclusion Criteria:

* Adults 25-70 years old
* Moderate-severe OSA (AHI 15+)
* First prescription of CPAP therapy
* Undiagnosed HBP
* Smartphone use and technological skills
* Informed consent

Exclusion Criteria:

* Antihypertensive drug
* Cardiovascular comorbidity: atrial fibrilation, heart failure, ischemic heart disease, stroke
* Reduced perfusion (e.g. Raynaud)
* Severe/Advanced chronic disease
* Central apnea
* Pregnancy
* Shift work
* Other social issues: misunderstanding/miscommunication

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the AKTIIA OBPM systolic blood pressure (SBP) at 12 weeks | 1 week pre-CPAP and 1 week post-CPAP at the end of 12 weeks AKTIIA OBPM
  Change in 24h/7d average SBP from week 0 (pre-CPAP) to week 12 (post-CPAP). SBP expressed in mmHg (millimeters of mercury)

SECONDARY OUTCOMES:
Change from baseline in the left ventricular global longitudinal strain (LV-GLS) at 12 weeks | Baseline prep-CPAP and at the end of 12 weeks AKTIIA OBPM
  Change in LV-GLS from pre-CPAP speckle tracking echocardiography (STE) to post-CPAP STE at week 12 (post-CPAP). LV-GLS values are reported as absolute numbers. By convention, GLS is expressed as a negative number (normal range, -19% to -20%), and more negative LV GLS values represent better systolic performance.

OTHER OUTCOMES:
Change from OSA diagnosis in Epworth Sleepiness Scale scoring at 12 weeks | Baseline at OSA diagnosis (pre-CPAP) and at the end of 12 weeks AKTIIA OBPM (post-CPAP)
  Change in ESS scoring from OSA diagnosis (pre-CPAP) to ESS scoring at the end of 12 weeks (post-CPAP). The ESS score is based on 8 questions and a scale of 0 to 24. The scale estimates whether the participants are experiencing excessive sleepiness due to OSA and its improvement with CPAP therapy. A normal score (no diurnal sleepiness) is less than 11 points.
Usability of AKTIIA system and Patient Experience with AKTIIA OBPM at 12 weeks | At the end of 12 weeks AKTIIA OBPM
  Participants answer an anonymous survey of several questions about the usability of the AKTIIA system and their experience and opinion about continuous blood pressure monitoring for 12 weeks. The questions are asked on a Likert scale from 1 to 5, with 5 being the best satisfaction/opinion.

CONTACTS AND LOCATIONS:
Overall Officials: Mikel Azpiazu, MD, Principal Investigator — Hospital Universitario Araba
Locations (1):
- Hospital Universitario Araba, Vitoria-Gasteiz, Araba, Spain

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 1 month after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Data obtained through this study may be provided to qualified researchers with academic interest in sleep apnea, HBP or AKTIIA OBPM. Data or samples shared will be coded, with no protected health information included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
  Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact to migueljavier.azpiazublocona@osakidetza.eus

REFERENCES:
- [Background] Sola J, Cortes M, Perruchoud D, De Marco B, Lobo MD, Pellaton C, Wuerzner G, Fisher NDL, Shah J. Guidance for the Interpretation of Continual Cuffless Blood Pressure Data for the Diagnosis and Management of Hypertension. Front Med Technol. 2022 May 17;4:899143. doi: 10.3389/fmedt.2022.899143. eCollection 2022. PMID 35655524
- [Background] Tadic M, Gherbesi E, Faggiano A, Sala C, Carugo S, Cuspidi C. The impact of continuous positive airway pressure on cardiac mechanics: Findings from a meta-analysis of echocardiographic studies. J Clin Hypertens (Greenwich). 2022 Jul;24(7):795-803. doi: 10.1111/jch.14488. Epub 2022 Jun 13. PMID 35695237
- [Background] Bazzano LA, Khan Z, Reynolds K, He J. Effect of nocturnal nasal continuous positive airway pressure on blood pressure in obstructive sleep apnea. Hypertension. 2007 Aug;50(2):417-23. doi: 10.1161/HYPERTENSIONAHA.106.085175. Epub 2007 Jun 4. PMID 17548722
- [Background] Bradley TD, Floras JS. Obstructive sleep apnoea and its cardiovascular consequences. Lancet. 2009 Jan 3;373(9657):82-93. doi: 10.1016/S0140-6736(08)61622-0. Epub 2008 Dec 26. PMID 19101028

DOCUMENTS (2):
  • Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT06446934/SAP_000.pdf
  • Informed Consent Form (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT06446934/ICF_001.pdf